CLINICAL TRIAL: NCT00066157
Title: Alzheimer's Disease: Therapeutic Potential of Estrogen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001-477; R01AG017196-03 (NIH); FDA IRB approval M1285; NIH grant AG17196-03; IA0048 (Other: Study Team)
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Hormone replacement therapy; Postmenopausal women
MeSH Terms: conditions — Alzheimer Disease | interventions — Estrogen Replacement Therapy; Medroxyprogesterone; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): estradiol patch and medroxyprogesterone
  Interventions: Drug: Transdermal estradiol; Drug: Medroxyprogesterone
- 2 (Active Comparator): estradiol patch and placebo pill
  Interventions: Drug: Transdermal estradiol; Drug: Placebo
- 3 (Active Comparator): placebo patch and medroxyprogesterone
  Interventions: Drug: Medroxyprogesterone; Drug: Placebo Patch
- 4 (Placebo Comparator): placebo patch and placebo pill
  Interventions: Drug: Placebo Patch; Drug: Placebo

INTERVENTIONS:
Drug: Transdermal estradiol — 50 micrograms (low-dose) or 100 micrograms (high-dose) transdermal 17-ß-estradiol patch, changed every 3 days, for 12 months
  Other Names: 17 (beta) estradiol transdermal patch; Estrogen replacement therapy
  Arms: 1; 2
Drug: Medroxyprogesterone — 2.5mg tablet daily for 12 months
  Other Names: progesterone
  Arms: 1; 3
Drug: Placebo Patch — Transdermal placebo patch, changed every 3 days, for 12 months
  Arms: 3; 4
Drug: Placebo — Placebo tablet daily for 12 months
  Arms: 2; 4

SUMMARY:
This is a 15-month study to determine the effectiveness of hormone replacement therapy in improving memory and the ability to live independently in postmenopausal women with Alzheimer's disease.

DETAILED DESCRIPTION:
Estrogen is a naturally occurring hormone produced in a woman's body. The purpose of this 15-month study is to determine the effectiveness of hormone replacement therapy in improving memory and the ability to live independently in postmenopausal women with Alzheimer's disease and without other dementias.

Patients who volunteer for this study will either receive a patch containing 17-ß-estradiol or will receive an inactive placebo patch. In addition, patients will be given either medroxyprogesterone or an inactive placebo pill. Neither the volunteers nor the study staff will know which type of patch or pill a patient receives. Patients must be generally healthy and have mild-to-moderate dementia. There must be a patient caregiver who can watch for side effects and ensure that the patient takes the study medications on schedule. Patients will undergo neuropsychological tests and an evaluation of the ability to live independently at each visit as well as laboratory evaluations, such as the taking of blood. Each visit will last approximately 3 hours. A total of 160 participants are being recruited.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with Alzheimer's disease and without other dementias (diagnosed by study staff or from an outside clinic)
* Mini Mental State Examination score greater than 15/30

Exclusion Criteria:

* History of cancer of reproductive tissues
* History of deep vein thrombosis or blot clots
* Diabetes
* Heart disease or stroke
* Liver problems including hepatitis
* Severe vision or hearing problems
* Tobacco use
* Lack of an adequate caregiver
* inability to perform psychometric testing

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cognition: delayed recall on Buschke Selective Reminding Test; Stroop Interference condition--completion time and errors; Clinician-rated Interview Based Impression of Change | Baseline and 1, 3, 6, 12, and 15 months

SECONDARY OUTCOMES:
Skills of Independent Living: Physical functioning Performance (PFP) | Baseline and 1, 3, 6, 12, and 15 months
Bioassays (Estradiol, estrone, medroxyprogesterone, FSH, influence of ApoE genotype in responsivity to estrogen) | Baseline and 1, 3, 6, 12, and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Asthana, MD, Principal Investigator — University of Wisconsin - Madison, William S. Middleton VA Hospital
Locations (1):
- University of Wisconsin Memory Research Program, Madison, Wisconsin, United States

REFERENCES:
- [Background] Cholerton B, Gleason CE, Baker LD, Asthana S. Estrogen and Alzheimer's disease: the story so far. Drugs Aging. 2002;19(6):405-27. doi: 10.2165/00002512-200219060-00002. PMID 12149049
- [Background] Asthana S, Baker LD, Craft S, Stanczyk FZ, Veith RC, Raskind MA, Plymate SR. High-dose estradiol improves cognition for women with AD: results of a randomized study. Neurology. 2001 Aug 28;57(4):605-12. doi: 10.1212/wnl.57.4.605. PMID 11524467
- [Background] Asthana S, Craft S, Baker LD, Raskind MA, Birnbaum RS, Lofgreen CP, Veith RC, Plymate SR. Cognitive and neuroendocrine response to transdermal estrogen in postmenopausal women with Alzheimer's disease: results of a placebo-controlled, double-blind, pilot study. Psychoneuroendocrinology. 1999 Aug;24(6):657-77. doi: 10.1016/s0306-4530(99)00020-7. PMID 10399774